CLINICAL TRIAL: NCT03115840
Title: Long-term Outcomes of Physical Activity in Older Adults With Critical Illness
Brief Title: Measuring Outcomes of Activity in Intensive Care
Acronym: MOSAIC
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Wes Ely, Professor of Medicine, Allergy/Pulmonary & Critical Care, Vanderbilt University Medical Center
Other Study IDs: 116157; 1K76AG054864-01 (NIH)
Record Dates: First submitted 2017-03-28; First posted 2017-04-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Critical Illness; Sepsis; Mechanical Ventilation; Physical Activity; Disability Physical; Muscle Weakness; Cognitive Impairment
MeSH Terms: conditions — Critical Illness; Sepsis; Motor Activity; Muscle Weakness; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults (≥18 years old) with critical illness

SUMMARY:
Millions of older adults are hospitalized for a critical illness each year and although they are more likely than ever to survive this illness, they commonly face significant morbidity in the form of disabilities in basic self-care activities and in mobility in the months and years afterwards. A better understanding of the underlying risk factors for disability following critical illness is greatly needed, including the effect that activity during hospitalization may have on these outcomes. Therefore, we designed the Measuring OutcomeS of Activity in Intensive Care (MOSAIC) observational study to evaluate the relationship between activity (measured more rigorously than in prior investigations) and disability, physical function, and cognitive function in survivors of critical illness 3 and 12 months after ICU discharge.

DETAILED DESCRIPTION:
The MOSAIC observational study will measure activity in critically ill patients for up to 28 days in the hospital using two different, objective measures, a clinical mobility scale and accelerometry. We will evaluate the independent association between activity and outcomes 3 and 12 months after ICU discharge. Specifically, Aim 1 will determine the relationship between activity and disability in ADLs and mobility. Aim 2a will determine the relationship between activity and physical and cognitive function. Aim 2b will evaluate physical and cognitive function as mediators of long-term disability. Aim 3a will determine the relationship between activity and biomarkers of inflammation and coagulation. Aim 3b will determine the relationship between these biomarkers of inflammation and coagulation and disability, physical and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients (≥18 years old),
2. in a medical or surgical ICU at Vanderbilt University Medical Center or The Ohio State University Medical Center, and
3. are being treated for respiratory failure or shock.

Exclusion Criteria:

1. Rapidly resolving organ failure criteria, indicated by planned immediate discontinuation of mechanical ventilation, NIPPV, and/or vasopressors at the time of screening for study enrollment, such that the patient will no longer meet inclusion criteria.
2. Cumulative hospital days (ICU plus non-ICU) of five or greater in the last 30 days prior to meeting all inclusion criteria.
3. Inability to live independently at baseline due to acquired or congenital disabling, physical, cognitive or mental health disorder requiring institutionalization (e.g., nursing home, skilled nursing facility, group home, long-term acute care hospital, rehab facility) or any patient who resides outside an institution with an inability to walk without the assistance of another person (e.g., patients with quadriplegia, paraplegia, double amputees, those with residual paralysis from stroke).
4. Acute or subacute severe neurologic (e.g., stroke anoxic injury, spinal cord injury) that is expected to prevent the patient from living independently after hospital discharge.
5. Body mass index >50
6. Active substance abuse or psychotic disorder (e.g., schizophrenia or schizo-affective disorder), recent (within the past 6 months) serious suicidal gesture necessitating hospitalization
7. Blindness, deafness, or inability to understand English that will preclude follow-up evaluation. Patients with laryngectomies and those with hearing impairments are eligible for enrollment if their medical condition permits them to communicate with research staff.
8. Expected death within 24 hours of enrollment or lack of commitment to aggressive treatment by family or the medical team (e.g., likely to withdraw life support measures within 24 hours of screening).
9. Prisoners
10. Patients who live further than 200 miles from an enrolling center and who do not regularly visit the area.
11. Patients who are homeless and have no secondary contact person available
12. Current enrollment in a study that does not allow co-enrollment
13. Inability to obtain informed consent from the patient or an authorized representative within 72 hours of meeting all inclusion criteria for the following reasons:

    1. Attending physician refusal
    2. Patient and/or surrogate refusal
    3. 72-hour period of eligibility was exceeded before the patient was screened
    4. Patient unable to consent and no surrogate available within 72 hours of meeting all inclusion criteria
14. Confirmed or suspected COVID-19 per local guidelines at the time of screen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with medical or surgical critical illness
Sampling Method: Non-Probability Sample
Enrollment: 312 (Estimated)
Dates: Start 2017-03-27 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Precipitating Events Project Disability Questionnaire | 12 months
  Questionnaire assessment of activities of daily living and mobility
Life Space Assessment Questionnaire | 12 months
  Questionnaire assessment of activities of community mobility

SECONDARY OUTCOMES:
Precipitating Events Project Disability Questionnaire | 3 months
  Questionnaire assessment of activities of daily living and mobility
Life Space Assessment Questionnaire | 3 months
  Questionnaire assessment of activities of community mobility
Survival | 30, 90, and 365 days
  Proportion of patients surviving at 30, 90, and 365 days
Ventilator-free days | out of 28 days
  Days alive and free of mechanical ventilation
Delirium and coma-free days | out of 28 days
  Days alive and without delirium or coma
ICU Length of Stay | up to 28 days
  Days spent in the ICU during the index hospitalization
Hospital Length of Stay | up to 28 days
  Days spent in the hospital during the index hospitalization
Short Physical Performance Battery | 3 months
  Performance Measure of Physical Function
Short Physical Performance Battery | 12 months
  Performance Measure of Physical Function
Handgrip Dynamometry | 3 months
  Performance Measure of Muscle Strength
Handgrip Dynamometry | 12 months
  Performance Measure of Muscle Strength
Repeatable Battery for the Assessment of Neuropsychological Status | 3 months
  Test of Global Cognition
Repeatable Battery for the Assessment of Neuropsychological Status | 12 months
  Test of Global Cognition
Trail Making Test Parts A & B | 3 months
  Test of Executive Function
Trail Making Test Parts A & B | 12 months
  Test of Executive Function

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Ohio State University Medical Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brummel NE, Balas MC, Morandi A, Ferrante LE, Gill TM, Ely EW. Understanding and reducing disability in older adults following critical illness. Crit Care Med. 2015 Jun;43(6):1265-75. doi: 10.1097/CCM.0000000000000924. PMID 25756418
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Gill TM, Allore HG, Gahbauer EA, Murphy TE. Change in disability after hospitalization or restricted activity in older persons. JAMA. 2010 Nov 3;304(17):1919-28. doi: 10.1001/jama.2010.1568. PMID 21045098